CLINICAL TRIAL: NCT00709982
Title: An Open-label Pharmacokinetic Drug Interaction Study of Folic Acid and 250 Mcg NGM/35 Mcg EE (ORTHO-CYCLEN) in Healthy Women..
Brief Title: A Drug Interaction Study of Folic Acid and Oral Contraceptive Tablets Containing Norgestimate (NGM) /Ethinyl Estradiol (EE) in Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR002380
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Drug Interactions; Healthy; Pharmacokinetics
Keywords: Norgestimate; Contraceptives, Oral; Ortho-Cyclen; Folic Acid; Ethinyl Estradiol
MeSH Terms: interventions — norgestimate; Ethinyl Estradiol; Folic Acid

INTERVENTIONS:
Drug: Norgestimate; Ethinyl Estradiol; Folic acid

SUMMARY:
The purpose of the study is to assess the effect of folic acid administration on the blood level and the breakdown products of OC study drug (250 mcg norgestimate[NGM]/35 mcg Ethinyl Estradiol [EE]) tablets. The effect of study drug tablet intake on the blood level of folic acid is also determined.

DETAILED DESCRIPTION:
This is a single-center, open-label, pharmacokinetic drug interaction study between folic acid (1 mg) and study drug (250 mcg NGM/35 mcg EE) in 2 groups of at least 20 healthy women each. In Group 1, a single oral dose of 250 mcg NGM/35 mcg EE study drug was administered to the healthy volunteers at the study site on Days 1 and 17 and folic acid 1 mg was administered orally on Days 4 to 18; in Group 2, folic acid 1 mg was administered orally on Days 1 and 17 at the study site and 1 tablet of study drug was administered on Days 2 to 17. Blood samples were collected at specified times for 72 hours postdose on Days 1 and 17 for the healthy volunteers in Group 1 for determination of blood levels of norelgestromin (NGMN), and norgestrel (NG) [the active breakdown product of NGM], and EE. For the healthy volunteers in Group 2, blood samples were collected for 24 hours after the folic acid dose on Days 1 and 17 for determination of plasma levels of total folates. Safety was evaluated based on the following: the incidence, type and severity of adverse events; clinical laboratory tests; vital sign and electrocardiogram (ECGs) measurements; and physical examinations. Oral temperature, pulse, respiratory rate, and sitting blood pressure (BP) were taken before dosing on Days 1 and 17. For Group 1, measurements were taken before and at least 15 minutes after the 24-hour (Days 2 and 18), 48-hour (Days 3 and 19), and 72-hour (Day 4) pharmacokinetic blood draw; and at study completion (Day 20) or early withdrawal. For Group 2, measurements were taken before and at least 15 minutes after the 24-hour pharmacokinetic blood draw on Days 2 and 18; and at study completion (Day 18) or early withdrawal. Physical and gynecologic examinations and 12-lead ECGs were performed at screening and at study completion or early withdrawal. Blood samples for blood chemistry, hematology, and urine samples for urinalysis were collected at the screening visit and at the follow-up visit or early withdrawal.

Oral contraceptives tablet (250 mcg NGM/35 mcg EE); Folic acid tablet (1 mg). In Group 1, a single oral dose of (250 mcg NGM/35 mcg EE) study drug was administered on Days 1 and 17 and folic acid 1 mg was administered orally on Days 4 to 18; in Group 2, folic acid 1 mg was administered orally on Days 1 and 17 and 1 tablet of study drug was administered on Days 2 to 17. Study drugs were taken with 240 mL (8 oz) of water at approximately 8:00 a.m.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonpregnant, nonlactating, nonsmoking women, weighing at least 110 pounds
* With regular menstrual cycles
* A body mass index between 16 and 29.9 kg/m2
* And having a hematocrit of at least 36%

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to sex hormonal therapy including: thromboembolic disorders' cerebral vascular or coronary artery disease, chronic untreated hypertension, or migraines, benign or malignant liver tumor that developed during the use of OC
* Known or suspected estrogen-dependent neoplasia
* Presence of disorders commonly accepted as contraindications to combined OC including: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, or liver disease
* Intake any multivitamin or folic acid-containing supplements within 21 days before study admission
* Used a steroid hormone-containing intrauterine device within 3 months before study admission
* Used any medications that were known cytochrome P-450 enzyme inducers or inhibitors (e.g., St. John's Wort, cimetidine or rifampin), within 60 days before dosing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2005-05; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetic drug interaction between folic acid and the study drug (250 mcg NGM and 35 mcg EE) as measured by the pharmacokinetics of the active breakdown product of NGM, norelgestromin (NGMN), and EE.

SECONDARY OUTCOMES:
Measure the pharmacokinetics of the active metabolite of NGM, norgestrel (NG). Evaluate the effect of the study drug on the pharmacokinetics of folic acid. Assess the safety.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A drug interaction study of folic acid and oral contraceptive tablets containing norgestimate (250 mcg)/ethinyl estradiol (35 mcg) in healthy women — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=475&filename=CR002380_CSR.pdf